CLINICAL TRIAL: NCT05338827
Title: Comparison of a Polyvinyl Chloride Tube With a Wire-reinforced Tube for Tracheal Intubation Through the SaCoVLM Video Laryngeal Mask Airway: a Randomized Controlled Study
Brief Title: Comparison of a Polyvinyl Chloride Tube With a Wire-reinforced Tube for Tracheal Intubation Through the SaCoVLM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Yongtao Sun, Professor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: SaCoVLM
Record Dates: First submitted 2022-04-14; First posted 2022-04-21 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Laparoscopic Surgery
Keywords: SaCO Video Laryngeal Mask Airway; intubating laryngeal mask airway; laryngeal mask airway; supraglottic airway devices; endotracheal intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Polyvinyl Chloride Tube group (Experimental): The PVC tube used is a stiff tube with an anterior curvature of approximately 130°, which retains the additional curvature imposed by its passage through the ventilation conduit of the ILMA. The SaCoVLM glottic exposure grade was referred to the endoscopic view grading system. If the SaCoVLM glottic exposure grade is 1 or 2, a lubricated tracheal tube will be inserted in a conventional manner with the curvature of the tracheal tube aligned along the intrinsic curvature of the SaCoVLM. The passage of the tracheal tube into the glottis will be visualised. If there is a discrepancy in the alignment of the tracheal tube exiting from the SaCoVLM and the glottis that will prevent the passage of the tracheal tube into the glottis, the tracheal tube will be withdrawn and manipulations (rotation of the tracheal tube or up/down manoeuvre) will be performed in an attempt to align the glottis and tracheal tube tip to facilitate intubation. Such manoeuvres, if performed, will be recorded.
  Interventions: Procedure: Polyvinyl Chloride Tube group
- Wire-Reinforced Tube group (Experimental): In contrast to the PVC tube, the WR tube is flexible with a slightly anterior curvature. The SaCoVLM glottic exposure grade was referred to the endoscopic view grading system. If the SaCoVLM glottic exposure grade is 1 or 2, a lubricated tracheal tube will be inserted in a conventional manner with the curvature of the tracheal tube aligned along the intrinsic curvature of the SaCoVLM. The passage of the tracheal tube into the glottis will be visualised. If there is a discrepancy in the alignment of the tracheal tube exiting from the SaCoVLM and the glottis that will prevent the passage of the tracheal tube into the glottis, the tracheal tube will be withdrawn and manipulations (rotation of the tracheal tube or up/down manoeuvre) will be performed in an attempt to align the glottis and tracheal tube tip to facilitate intubation. Such manoeuvres, if performed, will be recorded.
  Interventions: Procedure: Wire-Reinforced Tube group

INTERVENTIONS:
Procedure: Polyvinyl Chloride Tube group — The anaesthesiologist will perform a visual screen for the SaCoVLM glottic exposure grade after the SaCoVLM is successfully inserted. The SaCoVLM glottic exposure grade was referred to the endoscopic view grading system. If the SaCoVLM glottic exposure grade is 1 or 2, a lubricated tracheal tube will be inserted in a conventional manner with the curvature of the tracheal tube aligned along the intrinsic curvature of the SaCoVLM. The passage of the tracheal tube into the glottis will be visualised. If there is a discrepancy in the alignment of the tracheal tube exiting from the SaCoVLM and the glottis that will prevent the passage of the tracheal tube into the glottis, the tracheal tube will be withdrawn and manipulations (rotation of the tracheal tube or up/down manoeuvre) will be performed in an attempt to align the glottis and tracheal tube tip to facilitate intubation. Such manoeuvres, if performed, will be recorded.
  Arms: Polyvinyl Chloride Tube group
Procedure: Wire-Reinforced Tube group — The anaesthesiologist will perform a visual screen for the SaCoVLM glottic exposure grade after the SaCoVLM is successfully inserted. The SaCoVLM glottic exposure grade was referred to the endoscopic view grading system. If the SaCoVLM glottic exposure grade is 1 or 2, a lubricated tracheal tube will be inserted in a conventional manner with the curvature of the tracheal tube aligned along the intrinsic curvature of the SaCoVLM. The passage of the tracheal tube into the glottis will be visualised. If there is a discrepancy in the alignment of the tracheal tube exiting from the SaCoVLM and the glottis that will prevent the passage of the tracheal tube into the glottis, the tracheal tube will be withdrawn and manipulations (rotation of the tracheal tube or up/down manoeuvre) will be performed in an attempt to align the glottis and tracheal tube tip to facilitate intubation. Such manoeuvres, if performed, will be recorded.
  Arms: Wire-Reinforced Tube group

SUMMARY:
To compare a polyvinyl chloride tube with a wire-reinforced tube for tracheal intubation through the SaCoVLM video laryngeal mask airway, to observe the success rate of intubation and the incidence of postoperative adverse reactions, and to explore the best type of endotracheal tube through the SaCoVLM video laryngeal mask airway, so as to provide reference for its clinical application.

DETAILED DESCRIPTION:
1. At present, there are few studies on intubation through SaCoVLM video laryngeal mask airway. It is proposed that endotracheal intubation through SaCoVLM video laryngeal mask airway is to verify its feasibility.
2. The purpose is to explore the best type of endotracheal tube by observing the success rate of intubation through SaCoVLM video laryngeal mask airway and the incidence of postoperative adverse reactions.
3. By observing the hemodynamic changes of the polyvinyl chloride tubes and the wire-reinforced tube during intubation through SaCoVLM video laryngeal mask airway , the effects of the two tracheal tubes on the hemodynamics of patients were compared.
4. By observing the optimized operation which can improve the success rate of tracheal intubation in the experiment, it can be better applied in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled to accept elective laparoscopic surgery under general anaesthesia.
2. Aged 18-70 years.
3. Body mass index (BMI) 18.5-27.9 kg/m2.
4. ASA class I-III.

Exclusion Criteria:

1. Neurological or psychiatric diseases (such as schizophrenia and depression), or unconscious.
2. Severe cardiopulmonary dysfunction.
3. Vocal cord injury, pharyngeal disease or history of neck surgery.
4. Risk of reflux aspiration and indwelling nasogastric tube before and after surgery.
5. Mouth opening less than 2 cm, limitation of cervical extension, modified Mallampati score IV.
6. SaCoVLM glottic exposure grade 3 or 4.
7. Participated in other clinical studies during the last 3 months.
8. Refused to give informed consent for the clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
The total success rate of tracheal intubation | From the beginning of the general anaesthesia induction to tracheal intubation through an SaCO Laryngeal Mask Airway. It will take up to half hour or 1 hour.
  defined as the cumulative third-attempt intubation success rate

SECONDARY OUTCOMES:
Successful insertion rate on the first attempt | From the beginning of the general anaesthesia induction to tracheal intubation through an SaCO Laryngeal Mask Airway. It will take up to 15 minutes or half hour.
  tracheal intubation is considered successful if the endotracheal tube slides through the LMA without any resistance, and tracheal intubation was confirmed by the laryngeal mask visual screen and detection of end-tidal carbon dioxide (CO2).
Time of tracheal intubation | From the beginning of the general anaesthesia induction to tracheal intubation through an SaCO Laryngeal Mask Airway. It will take up to 15 minutes or half hour.
  defined as the time from picking up the tracheal tube to the appearance of three standard end-tidal CO2 waveforms on the monitor.
Site of first contact of tracheal intubation | From the beginning of the general anaesthesia induction to tracheal intubation through an SaCO Laryngeal Mask Airway. It will take up to 15 minutes or half hour.
  which will be identified with the SaCoVLM visual screen (four areas are defined based on the glottic opening: the interarytenoid fold, the left and right aryepiglottic, the vestibular and vocal folds, and the tubercle of the epiglottis).8
Adjustment action for tracheal intubation | From the beginning of the general anaesthesia induction to tracheal intubation through an SaCO Laryngeal Mask Airway. It will take up to 15 minutes or half hour.
  if tracheal intubation is unsuccessful after the first attempt, the tube will be pulled 2 cm, rotated and then advanced. If this attempt is unsuccessful, the tube will again be pulled 2 cm, adjusted to the SaCoVLM by the up-down manoeuvre, rotated and then advanced. If tracheal intubation is accomplished after either manoeuvre, this is considered a success and the manoeuvre used would be documented.
Haemodynamic fluctuation | It will take up to half hour or 1 hour.
  the systolic and diastolic blood pressure, mean arterial pressure and HR after induction, immediately, and 3 min after insertion of the laryngeal mask; immediately and 3 min after tracheal intubation; 3 min before extubation; and immediately and 3 min after extubation are recorded.
Incidence of trauma as evidenced by blood | It will take up to half hour or 1 hour.
  incidence of trauma as evidenced by blood on ILMA or endotracheal tube after removal
Incidence rate of postoperative sore throat, hoarseness and dysphagia at 24 hours after the surgery | one day after the surgery.
  the severity of sore throat will be evaluated using a numerical rating scale (0=no sore throat, 10=worst sore throat imaginable). Hoarseness will be classified as mild, moderate or severe (overall dysphonia grade, roughness, breathiness, asthenia and strain score). Dysphagia will be classified as normal, mild, moderate or severe according to the severity.

CONTACTS AND LOCATIONS:
Overall Officials: Yongtao Sun, doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University
Locations (1):
- Yongtao Sun, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao Z, Guo Y, Gao X, Wang W, Zhang M, Liu MJ, Chen L, Liu Y, Zhang X, Sun Y, Wang Y. Comparison of a polyvinyl chloride tube with a wire-reinforced tube for tracheal intubation through the SaCoVLM video laryngeal mask airway: protocol for a randomised controlled study. BMJ Open. 2022 Dec 14;12(12):e066084. doi: 10.1136/bmjopen-2022-066084. PMID 36517088